CLINICAL TRIAL: NCT07243847
Title: Artificial Deep Learning-Based Model for Predicting Postoperative Recurrence in Gastric Cancer
Brief Title: Recurrence and Prognosis Prediction Model for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Lu, Clinical Professor, Fudan University
Other Study IDs: Prediction model(GC)
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer (GC)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: surgery and/or chemo — Deep learning model

SUMMARY:
This study, utilizing a large-scale multicenter Eastern database, has established a Deep Learning-based predictive model for recurrence following gastric cancer surgery, which demonstrates robust discriminatory power for early recurrence. Furthermore, the individualized recurrence probability generated by this model can predict long-term postoperative prognosis and effectively stratify patients based on risk, thereby guiding personalized treatment choices. This individualized risk probability is also applicable to both adjuvant chemotherapy and neoadjuvant chemotherapy populations, offering valuable support for precision treatment in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed gastric adenocarcinoma; No distant metastases confirmed by preoperative examinations such as chest X-ray, abdominal ultrasonography, and upper abdominal computed tomography; Achievement of R0 resection.

Exclusion Criteria:

Presence of distant metastases detected preoperatively or intraoperatively; Prior neoadjuvant chemotherapy or radiotherapy; Incomplete general clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective analysis was conducted on the clinicopathological data of patients who underwent radical gastrectomy for gastric cancer between 2001 and 2022 at 13 tertiary hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
recurrence | 3 year after surgery

IPD SHARING:
Plan to Share IPD: No